CLINICAL TRIAL: NCT04390789
Title: Outcome Following Single-visit And Multiple-visit Nonsurgical Endodontic Retreatment
Brief Title: Single And Multiple-visit Endodontic Retreatment Outcome.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Kajal Bhayani
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2019-12

CONDITIONS: Apical Periodontitis
Keywords: Nonsurgical Retreatment, Single Visit; Multi visit, Calcium Hydroxide; Outcome
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single visit retreatment (Experimental): nonsurgical root canal retreatment will be carried out in single visit.
  Interventions: Procedure: Non surgical Single visit Retreatment
- multi visit retreatment (Active Comparator): In this group,GP removal and biomechanical preparation will be carried out in first visit,after which calcium hydroxide dressing will be placed and temporarily restored.after 7 days,in second visit obturation will be done followed by permanent restoration
  Interventions: Procedure: Multi visit Retreatment with calcium hydroxide dressing

INTERVENTIONS:
Procedure: Non surgical Single visit Retreatment — Non-surgical endodontic retreatment will be carried out in single visit.
  Arms: single visit retreatment
Procedure: Multi visit Retreatment with calcium hydroxide dressing — In this group,GP removal and biomechanical preparation will be carried out in first visit,after which calcium hydroxide dressing will be placed and temporarily restored.after 7 days,in second visit obturation will be done followed by permanent restoration
  Arms: multi visit retreatment

SUMMARY:
This study will compare the outcome of single visit retreatment and multi-visit retreatment in cases of failed root canal treated teeth.

DETAILED DESCRIPTION:
Retreatment is defined as a procedure to remove root canal filling materials from the tooth, followed by cleaning, shaping and obturating the canals.Although initial root canal therapy has been shown to be a predictable procedure with a high degree of success, failures can occur after treatment. Recent publications have reported failure rates of 14%-16% for initial root canal treatment. In order to prevent tooth loss in such cases, nonsurgical retreatment or apical surgery is often indicated.

In this study subjects will be assigned to either the single-visit and multi-visit nonsurgical endodontic retreatment. The allocation will be performed once the chemomechanical preparation is completed.

Clinical and radiographic success rate will be considered as primary outcome. Follow up will be carried out every 3 months, till 12-month period.

Pain intensity will be considered as secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patient willingness to participate in the study.
* Previously root filled Permanent teeth with post-treatment apical periodontitis requiring nonsurgical root canal retreatment.
* Failure of previous root canal treatment will be determined based on clinical and radiographic findings. Clinical indicators of failure will include pain, tenderness to palpation/percussion, swelling, sinus tract.Radiographic criteria will include persistent periapical radiolucent lesions in teeth in which initial treatments were performed at least 4 years previously.
* Root canal fillings no more than 4mm short of the apex.
* Patients showing no significant systemic disease

Exclusion Criteria:

* Patients who are pregnant, diabetic, immunocompromised, serious medical illness or requiring antibiotic premedication.
* Patient under 18 years of age.
* Patient under corticosteroid use.
* Patients with history of antibiotic use in last 3 months or analgesic use in last one week will also be excluded.
* Multiple teeth that require treatment to eliminate the possibility of pain referral.Patients with unrestorable carious lesions, fractures involving the periodontium, and/or periodontal pockets ≥ 4mm deep or having marginal or furcal bone loss due to periodontitis .
* Teeth with the procedural errors preventing access to apical third and missed canals will be excluded.
* Teeth that are not suitable for rubber dam isolation.
* Teeth with intraradicular post.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-12-15 (Actual); Primary Completion 2020-06-15 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
Clinical and radiographic success | Baseline to 1 year
  Criteria of clinical success:
  Absence of pain and tenderness to palpation/ percussion, absence of sinus or any associated soft tissue swelling, tooth mobility of grade-I or less, and no deterioration in periodontal probing depth as compared with baseline measurements
  Criteria of radiographic Success:
  PAI score 1-Normal periapical structures, OR PAI Score 2-Small changes in bone structure.
  Criteria of radiographic Failure:
  PAI score 3-Changes in bone structure with some mineral loss, OR PAI Score 4-Apical periodontitis with well-defined radiolucent area, OR PAI Score 5-Severe periodontitis with exacerbating features

SECONDARY OUTCOMES:
Pain assessment | Baseline to 7days
  Visual analogue scale (VAS) from 0 to 10 will be used to record preoperative and post -operative pain.

CONTACTS AND LOCATIONS:
Overall Officials: Kajal Bhayani, Principal Investigator — POST GRADUATE INSTITUTE OF DENTAL SCIENCES, ROHTAK
Locations (2):
- India (2):
  - Post graduate institute of dental sciences, Rohtak, Haryana
  - Sanjay Tewari, Rohtak, Haryana

IPD SHARING:
Plan to Share IPD: No